CLINICAL TRIAL: NCT01590875
Title: Validation of the Durability of the Adenosine Effect in Verification of Pulmonary Vein Isolation
Brief Title: Validation Durability Adenosine Effect in Verification Pulmonary Vein Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Marcie G. Berger, MD, PI, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MCWPRO00016186
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation; pulmonary veins; adenosine
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adenosine arm (Experimental): 25 patients will be randomized to received 2 doses of adenosine 12 mg IV, 5 minutes apart after pulmonary vein isolation. During this time, will monitor for pulmonary vein reconnection, second dose of adenosine will be given only if no reconnection after initial dose.
  Interventions: Drug: Adenosine arm
- Observation arm (No Intervention): 25 patients will be randomized to 10 minute period of observation for pulmonary vein reconnection after documentation of pulmonary vein isolation. This will serve as the control arm.

INTERVENTIONS:
Drug: Adenosine arm — In the adenosine arm, 25 patients will be randomized to received 2 doses of adenosine 12 mg IV, 5 minutes apart after pulmonary vein isolation. During this time, will monitor for pulmonary vein reconnection, second dose of adenosine will be given only if no reconnection after initial dose. In the observation arm, 25 patients will be randomized to 10 minute period of observation for pulmonary vein reconnection after documentation of pulmonary vein isolation.
  Arms: Adenosine arm

SUMMARY:
Adenosine is used clinically to assess permanency of electrical isolation of pulmonary veins during atrial fibrillation ablation, however, the methodology has not been validated either in terms of the reproducibility of the adenosine response or the effect on clinical outcomes, namely whether using pulmonary vein reconnection to guide additional ablation lowers rate recurrent atrial fibrillation post ablation. Study will test the hypothesis that the response to adenosine used in this manner is reproducible over time.

DETAILED DESCRIPTION:
Patients undergoing pulmonary vein isolation as part of atrial fibrillation ablation will be randomized to treatment and control groups. Treatment group subjects will received 12 mg IV adenosine to evaluate pulmonary vein reconnection after initial electrical isolation is documented. If electrical reconnection is not observed at 5 minutes, a second dose of adenosine will be administered, monitoring again for electrical reconnection. Control patients will be observed for 10 minutes post initial electrical isolation of the pulmonary vein for spontaneous electrical reconnection. If reconnection is observed, veins will be re-isolated per standard clinical practice. This procedure will be repeated for each of a patient's pulmonary veins. Patients will be followed up at clinical visits to examine for adverse effects of procedure and/or adenosine administration as well as atrial fibrillation recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing atrial fibrillation ablation, pulmonary vein isolation by catheter for standard clinical indications

Exclusion Criteria:

* allergy or contraindication to adenosine,
* inability to give informed consent,
* currently taking dipyridamole,
* verapamil or theophylline and
* breast-feeding mothers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcie G Berger, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adenosine Arm | Observation Arm
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adenosine Arm | Observation Arm | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Full Range); unit: years] | 60 [50 to 70] | 60 [55 to 70] | 60 [50 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Vein Reconnection
Description: In treatment group, 30 minutes after all veins confirmed to be isolated with lasso catheter, 12 mg IV adenosine will be given to treatment group subjects, will monitor with lasso catheter for pulmonary vein reconnection for 5 minutes after adenosine administration.
Time Frame: 5 minutes post infusion first dose adenosine
Measure: Count of Participants; unit: Participants
Arm/Group | Adenosine Arm | Observation Arm
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10
Statistical Analysis 1: Comparison: Adenosine Arm; Kappa statistics on per pulmonary vein basis were used to determine the probability of recovery, transient recovery or no recovery with second adenosine dose compared with probability of same response after first adenosine dose; Test type: Equivalence — Kappa statistics on per pulmonary vein basis were used to determine the probability of recovery, transient recovery or no recovery with second adenosine dose compared with probability of same response after first adenosine dose; p < 0.01, no relevant statistical analysis

2. Primary Outcome: Pulmonary Vein Reconnection
Description: In treatment group, 30 minutes after all veins confirmed to be isolated with lasso catheter, 12 mg IV adenosine will be given to treatment group subjects, will monitor with lasso catheter for pulmonary vein reconnection for 5 minutes, if no reconnection, a second dose adenosine will be given and will monitor for additional 5 minutes for pulmonary vein reconnection. Criteria for pulmonary vein reconnection will be recurrence of local pulmonary vein electrical recordings noted on lasso catheter located within the vein. Pulmonary vein isolation is defined as disappearance of all local intracardiac electrograms within a pulmonary vein recorded on a 10 electrode circular catheter or lasso catheter positioned within the vein.
Time Frame: Pulmonary vein reconnection will be monitored for 5 minutes post second dose of adenosine, or on average for 15 minutes after initial electrical isolation of the pulmonary vein.
Measure: Count of Participants; unit: Participants
Groups:
- Adenosine Arm: 10 patients were randomized to received 2 doses of adenosine 12 mg IV, 5 minutes apart after pulmonary vein isolation. During this time, we monitored for pulmonary vein reconnection, second dose of adenosine was given only if no reconnection after initial dose.
  Of these 10 patients, 3 patients were noted to have pulmonary vein reconnection post initial dose of adenosine in at least one pulmonary vein. No patient demonstrated pulmonary vein reconnection with second dose of adenosine.
- Observation Arm: 10 patients were randomized to 10 minute period of observation for pulmonary vein reconnection after documentation of pulmonary vein isolation. This served as the control arm.
  Of these 10 patients, none demonstrated pulmonary vein reconnection during the 10 minute period of observation.
Arm/Group | Adenosine Arm | Observation Arm
Number analyzed (Participants) | 10 | 10
Participants
  Patients with PV reconnection | 3 | 0
  Patients without PV reconnection | 7 | 10
Statistical Analysis 1: Comparison: Adenosine Arm; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.01, kappa statistic

ADVERSE EVENTS:
Time Frame: Adenosine the drug administered in the study is short acting with half life of less than 10 seconds. Adverse event data was collected from the time of the first adenosine administration to 30 minutes after the final adenosine administration. Thus total time over which adverse event data were collected was approximately 45 minutes.
Groups:
- Adenosine Arm: 10 patients were randomized to received 2 doses of adenosine 12 mg IV, 5 minutes apart after pulmonary vein isolation. During this time, we monitored for pulmonary vein reconnection, second dose of adenosine was given to the 7 patients without reconnection after initial dose.
- Observation Arm: 10 patients were be randomized to 10 minute period of observation for pulmonary vein reconnection after documentation of pulmonary vein isolation. This served as the control arm.
Arm/Group | Adenosine Arm | Observation Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No